CLINICAL TRIAL: NCT00661024
Title: Randomized Clinical Trial Evaluating Visualization Versus Intraoperative Neuromonitoring of the Recurrent Laryngeal Nerves in Thyroid Surgery
Brief Title: Visualization Versus Intraoperative Neuromonitoring of the Recurrent Laryngeal Nerves in Thyroid Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Marcin Barczynski, MD, PhD, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BBN/501/ZKL/L
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Last update posted 2008-04-18 (Estimated); Status verified 2008-04

CONDITIONS: Thyroid Surgery
Keywords: thyroid surgery; recurrent laryngeal nerves visualization; intraoperative neuromonitoring; predictive values

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): RLN visualization alone
  Interventions: Procedure: intraoperative RLN visualization
- 2 (Experimental): IONM of the RLN
  Interventions: Procedure: intraoperative neuromonitoring of the RLN

INTERVENTIONS:
Procedure: intraoperative RLN visualization — intraoperative RLN visualization
  Other Names: V-G
  Arms: 1
Procedure: intraoperative neuromonitoring of the RLN — IONM
  Other Names: IONM-G
  Arms: 2

SUMMARY:
Some recent studies have shown that intraoperative neuromonitoring (IONM) can aid the recurrent laryngeal nerve (RLN) identification during thyroid surgery. However, the role of IONM in reducing the incidence of RLN injury rate and the value of this method in predicting postoperative RLN function remain controversial. Only a few published series represent level III of evidence and grade C of recommendation according to the evidence-based criteria (Sackett's classification, modified by Heinrich). Thus, the aim of this randomized clinical trial was to compare the impact of RLN visualization versus IONM on their morbidity following thyroid surgery.

DETAILED DESCRIPTION:
Apart from hypoparathyroidism, dysfunction of the recurrent laryngeal nerve (RLN) is the most common complication following thyroid surgery. In consequence, the voice impairment leading to communication work-related problems and affecting psychological and social aspects of the individual's functioning diminishes the overall quality of life, being the common reason for medicolegal claims and litigation. The reported RLN palsy rate varies in the literature from 0% (for first-time thyroid surgery performed by an experienced endocrine surgeon) to as much as 20% (for reoperative thyroid surgery or thyroid malignancy surgery performed in low-volume centers), depending mostly on the type of thyroid disease (benign vs. malignant goiter), type (first-time vs. reoperation) and the extent of thyroid resection (subtotal vs. total thyroidectomy), surgical technique (with or without routine RLN identification) and the surgeon's experience (low-volume vs. high-volume thyroid surgery center.

In 1938, Lahey from Boston reported a significantly lower incidence of RLN injuries following thyroidectomy with dissection and visualization of the nerves as compared to operations without nerve identification. Since that time, many prospective studies have confirmed this observation, advocating routine RLN identification as the gold standard in safe thyroid surgery. But even in the most experienced hands RLN palsy occurs occasionally, with an average frequency below 1% of nerves at risk due to variability in RLNs anatomy and difficulties in nerve identification by visual or palpation control in challenging conditions (e.g. advanced thyroid malignancy or reoperative thyroid surgery). On the other hand, the use of intraoperative electrical stimulation for identifying the RLN nerve was described in 1966. However, the technique of intraoperative neuromonitoring (IONM) of RLN did not gain any widespread popularity until the late nineties of the last century, when several commercial user-friendly systems based on electromyographic signal recording became available. In these IONM systems, the RLN nerve stimulation is registered by elicited laryngeal muscles activity through the endoscopic insertion of the electrodes into the vocal cords, open insertion of the needle electrodes into the vocal muscles through the cricothyroid ligament or with the use of endotracheal tube surface electrodes. In addition to a plethora of signal acquisition techniques used in IONM, there is no consensus regarding the optimal method for nerve activity recording (continuous recording of spontaneous nerve activity versus repetitive stimulation) and no agreement as to which quantitative electromyographic parameter should be used as a predictor of postoperative vocal cord dysfunction (supramaximal versus minimal stimulation of the nerve at the end of the operation).

Some recent studies have shown that IONM can aid the RLN identification. However, the role of IONM in reducing the incidence of RLN injury rate and the value of this method in predicting postoperative RLN function remain controversial. Only a few published series represent level III of evidence and grade C of recommendation according to the evidence-based criteria (Sackett's classification, modified by Heinrich). Large, prospective, randomized trials addressing these issues and allowing for grade A recommendations are lacking due to some ethical concerns and large numbers of patients in each arm (more than 7000 patients) needed to reach the appropriate power of the study. To fulfill this gap in evidence, we designed a medium-size, single-center, prospective randomized study suitable for drawing more meaningful conclusions. Thus, the aim of this study was to compare the impact of RLN visualization versus IONM on their morbidity following thyroid surgery.

ELIGIBILITY:
Inclusion Criteria:

* thyroid pathology qualified for first-time bilateral neck surgery

Exclusion Criteria:

* previous thyroid or parathyroid surgery,
* unilateral thyroid pathology eligible for minimally invasive approach (MIVAT),
* mediastinal goiter,
* preoperatively diagnosed RLN palsy,
* pregnancy or lactation,
* age below 18 years,
* high-risk patients ASA 4 grade (American Society of Anesthesiology),
* and inability to comply with the scheduled follow-up protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2006-01; Primary Completion 2007-06 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
the incidence of the recurrent laryngeal nerve injury | on 2nd postoperative day and than at 1, 2, 4, 6 and 12 months postoperatively, if paresis was noted on first examination

SECONDARY OUTCOMES:
the IONM-added value to RLN identification | intraopreratively
the value of IONM in prediction of postoperative vocal cords function | intraoperative data compared with observation of vocal cords function postoperatively on the 2nd day postop

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Barczynski, MD, PhD, Principal Investigator — Jagiellonian University; Stanislaw Cichon, Prof, MD, Study Chair — Jagiellonian University; Aleksander Konturek, MD, PhD, Study Director — Jagiellonian University
Locations (1):
- Department of Endocrine Surgery, Jagiellonian University College of Medicine, Krakow, 37 Pradnicka Street, Poland

REFERENCES:
- [Background] Dralle H, Sekulla C, Lorenz K, Brauckhoff M, Machens A; German IONM Study Group. Intraoperative monitoring of the recurrent laryngeal nerve in thyroid surgery. World J Surg. 2008 Jul;32(7):1358-66. doi: 10.1007/s00268-008-9483-2. PMID 18305996
- [Background] Snyder SK, Hendricks JC. Intraoperative neurophysiology testing of the recurrent laryngeal nerve: plaudits and pitfalls. Surgery. 2005 Dec;138(6):1183-91; discussion 1191-2. doi: 10.1016/j.surg.2005.08.027. PMID 16360407
- [Background] Tomoda C, Hirokawa Y, Uruno T, Takamura Y, Ito Y, Miya A, Kobayashi K, Matsuzuka F, Kuma K, Miyauchi A. Sensitivity and specificity of intraoperative recurrent laryngeal nerve stimulation test for predicting vocal cord palsy after thyroid surgery. World J Surg. 2006 Jul;30(7):1230-3. doi: 10.1007/s00268-005-0351-z. PMID 16773263
- [Background] Barczynski M, Konturek A, Cichon S. [Value of the intraoperative neuromonitoring in surgery for thyroid cancer in identification and prognosis of function of the recurrent laryngeal nerves]. Endokrynol Pol. 2006 Jul-Aug;57(4):343-6. Polish. PMID 17006834
- [Background] Thomusch O, Sekulla C, Machens A, Neumann HJ, Timmermann W, Dralle H. Validity of intra-operative neuromonitoring signals in thyroid surgery. Langenbecks Arch Surg. 2004 Nov;389(6):499-503. doi: 10.1007/s00423-003-0444-9. Epub 2004 Jan 13. PMID 14722777
- [Derived] Barczynski M, Konturek A, Cichon S. Randomized clinical trial of visualization versus neuromonitoring of recurrent laryngeal nerves during thyroidectomy. Br J Surg. 2009 Mar;96(3):240-6. doi: 10.1002/bjs.6417. PMID 19177420